CLINICAL TRIAL: NCT01697852
Title: Cluster Randomised Trial to Compare Effectiveness of the Combined Use of Indoor Residual Spraying (IRS) and Long-lasting Insecticidal Nets (LLINs) to LLINs Alone for Malaria Prevention in Muleba District, Kagera Region, Tanzania
Brief Title: The Combined Use of Indoor Residual Spraying (IRS) and Long-lasting Insecticidal Nets (LLINs) for Malaria Prevention
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITDCVP54
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Malaria
Keywords: vector control; LLIN; IRS
MeSH Terms: conditions — Malaria | interventions — bendiocarb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLIN plus IRS (Experimental): LLIN by universal coverage campaign 2 rounds of indoor residual spraying with bendiocarb insecticide
  Interventions: Other: Indoor residual spraying with bendiocarb; Other: LLIN by universal coverage campaign
- LLIN only (Active Comparator): LLIN by universal coverage campaign
  Interventions: Other: LLIN by universal coverage campaign

INTERVENTIONS:
Other: Indoor residual spraying with bendiocarb — 2 rounds of indoor residual spraying with bendiocarb insecticide, 4 months apart
  Other Names: Ficam
  Arms: LLIN plus IRS
Other: LLIN by universal coverage campaign — Long lasting Insecticide treated mosquito net
  Other Names: Olyset nets

SUMMARY:
The study is a cluster randomised trial to compare the effectiveness of indoor residual spraying (IRS) combined with the use of long lasting insecticidal nets (LLINs) with the effectiveness of LLINs alone for preventing malaria infection and morbidity. The primary outcome measure is prevalence of parasitaemia and anaemia in children aged 0.5-10 years, measured in cross sectional surveys. Secondary outcomes include relative population density for each mosquito vector species, malaria transmission as measured by entomological inoculation rates (EIR) by mosquito vector species, monitoring of resistance markers including kdr, and user acceptability of LLINs compared with IRS.

Findings from this study are expected to inform decision making so that resource utilization can be optimised.

ELIGIBILITY:
Inclusion Criteria:

* resident in selected cluster (village)

Exclusion Criteria:

* Not resident in selected cluster (village)

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22300 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malarial infection in children 6 months to 10 years | 9 months post randomisation

SECONDARY OUTCOMES:
Moderate to severe anaemia in children under 5 years | 9 months post randomisation
Post-spraying prevalence of infection with malarial parasites in children 6 months to 10 years | 6 months post randomisation

OTHER OUTCOMES:
Entomological Innoculation Rate | Malaria season post randomisation(Average value during 6 months after randomisation)
Relative abundance of adult Anopheles mosquitoes by species | Malaria season post randomisation (Average value during 6 months after randomisation)
genotypic markers of insecticide resistance in malaria vector mosquitoes | Malaria season post randomisation (Average value during 6 months after randomisation)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rowland, PHD, Principal Investigator — London School of Hygiene and Tropical Medicine; Immo Kleinschmidt, PHD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- PAMVERC office, Muleba, Kagera, Tanzania

REFERENCES:
- [Background] Kleinschmidt I, Schwabe C, Shiva M, Segura JL, Sima V, Mabunda SJ, Coleman M. Combining indoor residual spraying and insecticide-treated net interventions. Am J Trop Med Hyg. 2009 Sep;81(3):519-24. PMID 19706925
- [Result] West PA, Protopopoff N, Rowland MW, Kirby MJ, Oxborough RM, Mosha FW, Malima R, Kleinschmidt I. Evaluation of a national universal coverage campaign of long-lasting insecticidal nets in a rural district in north-west Tanzania. Malar J. 2012 Aug 10;11:273. doi: 10.1186/1475-2875-11-273. PMID 22882836
- [Derived] West PA, Protopopoff N, Wright A, Kivaju Z, Tigererwa R, Mosha FW, Kisinza W, Rowland M, Kleinschmidt I. Enhanced protection against malaria by indoor residual spraying in addition to insecticide treated nets: is it dependent on transmission intensity or net usage? PLoS One. 2015 Mar 26;10(3):e0115661. doi: 10.1371/journal.pone.0115661. eCollection 2015. PMID 25811379
- [Derived] West PA, Protopopoff N, Wright A, Kivaju Z, Tigererwa R, Mosha FW, Kisinza W, Rowland M, Kleinschmidt I. Indoor residual spraying in combination with insecticide-treated nets compared to insecticide-treated nets alone for protection against malaria: a cluster randomised trial in Tanzania. PLoS Med. 2014 Apr 15;11(4):e1001630. doi: 10.1371/journal.pmed.1001630. eCollection 2014 Apr. PMID 24736370
- See also: Related Info — http://pamverc.org